CLINICAL TRIAL: NCT00943020
Title: The Effects of Supplementing Glutamine on the Gastric Emptying Time of a Preoperative Metabolic Conditioning Drink in Healthy Volunteers: a Randomized Crossover Pilot Study
Brief Title: Effects of Glutamine on Gastric Emptying
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Mr Dileep N Lobo, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 09026
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Starvation
Keywords: Dietary supplement; Carbohydrate loading; Healthy volunteers; Anaesthesia; Surgery; Glutamine
MeSH Terms: conditions — Starvation | interventions — Lipids; Glutamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nutricia PreOp + Lipid (Active Comparator): Nutricia PreOp + Lipid
  Interventions: Dietary Supplement: Nutricia PreOp nutritional supplement; Dietary Supplement: Lipid
- Nutrica PreOP + Glutamine (Active Comparator): Nutrica PreOP + Glutamine
  Interventions: Dietary Supplement: Nutricia PreOp nutritional supplement; Dietary Supplement: Glutamine
- Nutricia PreOP (Experimental): Nutricia PreOP: carbohydrate only drink
  Interventions: Dietary Supplement: Nutricia PreOp nutritional supplement

INTERVENTIONS:
Dietary Supplement: Nutricia PreOp nutritional supplement — nutritional supplement
Dietary Supplement: Lipid — Drink
  Arms: Nutricia PreOp + Lipid
Dietary Supplement: Glutamine — Drink
  Arms: Nutrica PreOP + Glutamine

SUMMARY:
Surgical patients are usually starved for 8 hours before operation in order to ensure the stomach is empty and thus reduce the chances of vomiting during the anaesthetic. Recent studies have shown that this period of starvation is harmful as it 'weakens' the body before operation. To avoid the harmful effects of starvation, patients are now given carbohydrate (sugar-containing) drinks 2 to 4 hours before surgery. These drinks have been shown to make patients feel better, reduce sickness after the anaesthetic/surgery and result in a quicker recovery from operation. The optimum time of giving these drinks to patients before operation is unknown. Previous studies have shown that the drinks empty from the stomach within 2 - 4 hours depending on their ingredients. The investigators would like to study the effects of adding protein and fat to these drinks on how quickly the drinks empty from the stomach. This study will investigate the hormone responses of the body following intake of 3 different drinks in order to determine the mechanisms that underlie the control of stomach emptying. This information will also allow us to improve the design of these drinks and this could help patients who undergo surgery who receive them.

DETAILED DESCRIPTION:
The eligibility criteria for this study are as follows:

Interested participants will be asked to attend a screening interview during which the study procedures/risks/benefits will be explained, followed by a brief history and physical examination. If deemed necessary by the study investigator, a 7ml sample of blood will be taken for screening purposes. The volunteer will be deemed eligible for the study once they have passed the screening visit and [when performed] had normal screening blood investigation results.

Each volunteer will be studied 3 times, the order of which will be determined randomly by computer. Participants will report for the study at the Division of GI Surgery (E-floor, West Block, Queen's Medical Centre), at 7:15am. On arrival the subject's height and weight will be recorded and 'drip needle' will will be placed in the back of the wrist. The hand will be rested in a hand-heater allowing venous blood to be sampled.

The subject will be randomly allocated to receive one of the three study drinks. At 7:50am baseline blood will be sampled (10ml [1.5 tablespoons] via the drip needle). At 8am the volunteers will drink the study drink. The rate of stomach emptying will be measured by using Gamma scintigraphy (a specialised medical camera). The drinks will have added a tracer substance that is visible on the camera and allows us to follow drink as it passes through the stomach into the bowels. Each 'picture' of the stomach lasts 20 seconds and we plan to take these every 20 minutes for 4 hours after intake of the drink. At 20 minute intervals (until 220 mins have elapsed) 7ml (1 tablespoon) of blood will be sampled via the drip needle. The final 10 ml blood sample will be taken at 240 minutes following which the drip needle will be removed and the volunteers will be allowed home. The subsequent two studies will be performed 7 days following the first study.

In total 95ml (a sixth of a pint) blood will be taken during each of the 3 crossover studies which will be separated by a period of 7 days (i.e. a total of 285 ml [half a pint] blood will be required from each volunteer).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian volunteers aged 18-60 years,
* BMI of 20-25 kg/m2,
* Able to give voluntary written informed consent to participate in the study,
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures.

Exclusion Criteria:

* Any history of acute or chronic illness,
* Smoking,
* Regular medication or substance abuse,
* Have taken part in any other clinical study within the previous 3 months.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time following supplementation of a standardised carbohydrate drink with glutamine. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N Lobo, FRCS, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre Biomedical Research Unit, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Awad S, Constantin-Teodosiu D, Macdonald IA, Lobo DN. Short-term starvation and mitochondrial dysfunction - a possible mechanism leading to postoperative insulin resistance. Clin Nutr. 2009 Oct;28(5):497-509. doi: 10.1016/j.clnu.2009.04.014. Epub 2009 May 17. PMID 19446932
- [Derived] Awad S, Blackshaw PE, Wright JW, Macdonald IA, Perkins AC, Lobo DN. A randomized crossover study of the effects of glutamine and lipid on the gastric emptying time of a preoperative carbohydrate drink. Clin Nutr. 2011 Apr;30(2):165-71. doi: 10.1016/j.clnu.2010.09.008. Epub 2010 Oct 23. PMID 20971535